CLINICAL TRIAL: NCT06961383
Title: A Double Blind, Randomized, Placebo Controlled Phase 2b Study to Evaluate the Safety and Clinical Efficacy of Treatment With the Autologous Cell Therapy Product, NG01, in Patients With Secondary Progressive Multiple Sclerosis
Brief Title: Study of NG01 Cell Therapy in Secondary Progressive Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroGenesis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NG01-P2b-SPMS-US
Record Dates: First submitted 2025-04-21; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: Secondary progressive multiple sclerosis; Multiple sclerosis; Autologous cell therapy
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CRO Monitors, Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 100x10^6 cells (Experimental): 15 participants with SPMS will receive 4 IT administrations of NG01 (100×10^6 cells), 3 months apart
  Interventions: Biological: NG01 - Autologous bone marrow derived human stromal cells
- 50x10^6 cells (Experimental): 15 participants with SPMS will receive 4 IT administrations of NG01 (50×10^6 cells), 3 months apart
  Interventions: Biological: NG01 - Autologous bone marrow derived human stromal cells
- Placebo (Placebo Comparator): 15 participants with SPMS will receive 4 IT administrations of placebo solution, 3 months apart
  Interventions: Other: Sodium Chloride 0.9%

INTERVENTIONS:
Biological: NG01 - Autologous bone marrow derived human stromal cells — NG01 is a cellular therapy product of autologous stromal cells derived from the bone marrow of multiple sclerosis (MS) patients. NG01 is provided as a cell suspension for intrathecal injection.
  Arms: 100x10^6 cells; 50x10^6 cells
Other: Sodium Chloride 0.9% — The placebo for use in the NG01 clinical trial is 0.9% Sodium Chloride Solution for Injection
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of repeated intrathecal (IT) injection of NG01, autologous bone marrow derived human stromal cells, in treating Secondary Progressive Multiple Sclerosis (SPMS), compared to placebo.

The study will assess the proportion of participants demonstrating improvement in walking ability, defined as a reduction in the average time to complete the Timed 25-Foot Walk (T25FW) at 6, 9, and 12 months compared to baseline. This will be analyzed by the mean change in walking speed across these time points. The study will also evaluate the incidence and nature of treatment-emergent adverse events (AEs).

Participants will receive intrathecal administrations of NG01, by lumbar puncture, and will be followed up for 6 months after their fourth administration.

DETAILED DESCRIPTION:
This is a multi-center, international Phase 2b, dose finding, randomized, double-blinded, placebo-controlled, three arm study, designed to assess the safety and efficacy of 4 IT administrations of NG01, compared to placebo, with a 4-month run-in period followed by a period of 9 months treatment with 6 months of follow-up, in patients with SPMS. Participants will continue to receive their customary MS treatment regimen at a stable dose.

The study will enroll 45 participants with secondary progressive multiple sclerosis (SPMS), randomized in a 1:1:1 ratio, to receive four intrathecal administrations-3 months apart over a 9-month period-of either high-dose NG01, low-dose NG01, or placebo. All participants will undergo clinical and safety assessments throughout the 9-month treatment period.

Upon completion of the 9-month treatment period, double-blind treatment and assessment period, participants will be followed clinically for an additional 6 months. The primary clinical outcome assessment and magnetic resonance imaging (MRI) acquisition for imaging assessments will occur post-treatment initiation (baseline).

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 65 years old.
2. Diagnosis of SPMS.
3. Documented EDSS worsening over the 2 years prior to study entry of ≥1 point for participants with EDSS <6.0 at screening, and ≥0.5 point for participants with EDSS ≥6.0 at screening, or a documented worsening of at least 20% in the T25FW. If documented T25fW or EDSS is not available, a written summary of the clinical evidence of disability worsening over the previous 2 years and retrospective assessment of EDSS score from data up to 2 years prior to screening, must be submitted for central review by adjudication committee.
4. EDSS at the screening visit from 3.5 to 6.5 at screening.
5. T25FW at the screening visit of from 8.0 to 25 seconds.

Exclusion Criteria:

1. Documented clinical relapse during the 24 months prior to enrollment and/or evidence of enhancing lesions on an MRI obtained at screening.
2. Pregnancy, breast feeding or women with childbearing potential without an acceptable form of contraception.
3. History of a general chronic handicapping/incapacitating disease other than MS.
4. Participants with clotting disorders
5. Participants unable to undergo an MRI scan.
6. Participants with uncontrolled hepatic disorders, renal or cardiovascular disease, or cancer.
7. Laboratory tests out of normal ranges considered by the investigator as clinically significant.
8. Participants with history or current alcohol abuse or drug addiction.
9. Untreated or uncontrolled psychiatric disorders, or positive suicidal risk assessed by Columbia-Suicide Severity Rating Scale (C-SSRS).
10. Participation in another research study involving an investigational product (IP) in the 90 days prior to inclusion, or planned use of another IP during the study duration.
11. Participants who have ever received NG01/MSCs treatment.
12. Participants who, in the opinion of the investigator, are unable to fully comprehend the consenting process or likely to be non-compliant with the study procedures or for whom long-term follow-up seems difficult to achieve.
13. Relapse occurring between screening and randomization.
14. Less than 6 months of the current disease-modifying therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Walking Ability | 12 months
  Proportion of participants who achieved improvement in walking ability over baseline by mean change in walking speed based on the Timed 25-Foot Walk (T25FW) test, averaged over visits at month-6, month-9 and month-12. Baseline is defined as the change in average timed walk compared to baseline (average timed walk at 6-, 9-, 12-months minus baseline < 0)
Incidence of Treatment-Emergent Adverse Events (AEs) | 15 months
  The occurrence of treatment-related AEs will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5 following enrollment, NG01 or placebo administrations (intrathecal), and during the 6 months of follow-up.

SECONDARY OUTCOMES:
Walking Speed | 12 months
  The change in walking speed will be assessed based on the average of two separate T25FW tests obtained during each study visit.
  The proportion of responders with 10, 15 or 20% improvement in walking speed will be assessed based on the average of two separate T25FW tests obtained during each study visit.
Neuroimaging Parameters - Change in T2-hyperintense Lesion | 12 months
  Change in T2-hyperintense lesion number and volume will be assessed by 3 tesla (3T) brain Magnetic Resonance Imaging (MRI) using automated volumetric analysis.
Neuroimaging Parameters - Change in T1-hypointense Lesion | 12 months
  Change in T1-hypointense lesion volume will be assessed by 3 tesla (3T) brain MRI using automated volumetric analysis.
Neuroimaging Parameters - Change in Brain and Thalamus | 12 months
  Change in whole brain and thalamic volume will be assessed by 3 tesla (3T) brain MRI using automated volumetric analysis
Efficacy - Finger Dexterity | 12 months
  Finger dexterity will be assessed by the 9-hole peg test (9HPT)
Quality of Life (QoL) | 12 months
  Quality of Life (QoL) will be assessed by 12-Item Short Form Survey (SF-12).
  Patients fill out a 12-question survey which is then scored by a clinician or researcher. The survey includes the following domains:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
Fatigue | 12 months
  Level of fatigue will be assessed by Modified Fatigue Impact Scale (MIFS-21). The scores are 0 (Never), 1(Rarely), 2 (Sometimes), 3 (Often), 4 (Almost always).
  Physical Subscale can range from 0 to 36. Cognitive Subscale can range from 0 to 40. Psychosocial Subscale can range from 0 to 8. The subscale scores are computed by adding raw scores on specific questions, in accordance with questionnaire instructions.
  Total MFIS Score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales.
Walking ability | 12 months
  Walking will be assessed by 12-item Multiple Sclerosis Walking Scale (MSWS-12). The original scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item. In a version 2, three items are scored 1-3, and nine items are scored 1-5.
Efficacy - Congnition | 12 months
  Cognitive assessment will be done using the Symbol Digit Modalities Test (SDMT)
Change in Disability | 12 months
  Proportion of participants with no increase in month-3 confirmed disability worsening (CDW) will be assessed by Expanded Disability Status Scale (EDSS). The EDSS ranges from 0 to 10. Scores are in half unit steps - 3, 3.5, 4 and so on. The greater the level of disability, the higher the score out of ten.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Miami Hospital & Clinics - Sylvester Comprehensive Cancer Center - Neurology, Miami, Florida, United States
- Hadassah University Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrou P, Gothelf Y, Argov Z, Gotkine M, Levy YS, Kassis I, Vaknin-Dembinsky A, Ben-Hur T, Offen D, Abramsky O, Melamed E, Karussis D. Safety and Clinical Effects of Mesenchymal Stem Cells Secreting Neurotrophic Factor Transplantation in Patients With Amyotrophic Lateral Sclerosis: Results of Phase 1/2 and 2a Clinical Trials. JAMA Neurol. 2016 Mar;73(3):337-44. doi: 10.1001/jamaneurol.2015.4321. PMID 26751635
- [Background] Petrou P, Kassis I, Ginzberg A, Halimi M, Yaghmour N, Abramsky O, Karussis D. Long-Term Clinical and Immunological Effects of Repeated Mesenchymal Stem Cell Injections in Patients With Progressive Forms of Multiple Sclerosis. Front Neurol. 2021 May 31;12:639315. doi: 10.3389/fneur.2021.639315. eCollection 2021. PMID 34135843
- [Background] Petrou P, Kassis I, Levin N, Paul F, Backner Y, Benoliel T, Oertel FC, Scheel M, Hallimi M, Yaghmour N, Hur TB, Ginzberg A, Levy Y, Abramsky O, Karussis D. Beneficial effects of autologous mesenchymal stem cell transplantation in active progressive multiple sclerosis. Brain. 2020 Dec 1;143(12):3574-3588. doi: 10.1093/brain/awaa333. PMID 33253391
- [Background] Petrou P, Kassis I, Yaghmour NE, Ginzberg A, Karussis D. A phase II clinical trial with repeated intrathecal injections of autologous mesenchymal stem cells in patients with amyotrophic lateral sclerosis. Front Biosci (Landmark Ed). 2021 Oct 30;26(10):693-706. doi: 10.52586/4980. PMID 34719198